CLINICAL TRIAL: NCT03016182
Title: Effect of Remote Ischemic Preconditioning on Pulmonary Injury in Cardic Surgery
Brief Title: Remote Ischemic Preconditioning on Pulmonary Injury in Cardic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Su Liu, Principal Investigator, Xuzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XYFY-2017-004
Record Dates: First submitted 2017-01-07; First posted 2017-01-10 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Lung Injury; Remote Ischemic Preconditioning
MeSH Terms: conditions — Lung Injury

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Preconditioning(RIPC) (Active Comparator): 3 cycles of 5-min upper limb ischemia and 5-min reperfusion using a blood-pressure cuff inflated to a pressure 200mmHg will be given to RIPC
  Interventions: Procedure: Remote Ischemic Preconditioning
- Control (Placebo Comparator): Control group without remote ischemic preconditioning
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning — RIPC will be induced during anesthesia by 3 cycles of 5-min upper limb ischemia and 5-min reperfusion using a blood-pressure cuff inflated to a pressure 200mmHg
  Other Names: RIPC
  Arms: Remote Ischemic Preconditioning(RIPC)
Procedure: Control — Control group witnout remote ischemic preconditioning
  Arms: Control

SUMMARY:
During cardiac surgery with cardiopulmonary bypass , pulmonary dysfunction remains to be a problem complicating the postoperative course of the patients.Remote ischemic preconditioning(RIPC) with transient upper limb ischemia/reperfusion is a novel, simple, cost-free,non-pharmacological and non-invasive strategy.Recent several trials suggested that RIPC could provide pulmonary protection by reducing serum biomarkers,however,whether the RIPC can improve the clinical outcomes in patients undergoing on-pump cardiac surgery,is still uncertain.

The study hypothesis is: remote ischemic preconditioning will provide lung-protective effect and improve clinical outcomes in patients undergoing cardic surgery.

DETAILED DESCRIPTION:
Remote ischemic preconditioning (RIPC) protocol will be induced during anesthesia by 3 cycles of 5-min upper limb ischemia and 5-min reperfusion using a blood pressure cuff inflated to a pressure 200mmHg

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing heart surgery on cardiopulmonary bypass
2. Patients aged 18 years to 80 years

Exclusion Criteria:

1. Inability to give informed consent
2. Preoperative severe impairment of respiratory function (arterial oxygen tension (PaO2) <60 mmHg or FEV1<50% predicted)
3. Prior receipt of chemotherapy or radiation therapy or immunotherapy
4. left ventricular ejection fraction less than 30%
5. preoperative use of inotropics or mechanical assist device
6. Patients with significant hepatic dysfunction (Prothrombin>2.0 ratio)
7. Patients with known renal failure with a GFR<30 mL/min/1.73 m2
8. recent myocardial infarction (within 7 days)
9. Systemic or local active infections (either clinically defined or suggested by evidence such as elevated C-reactive protein levels, leukocytosis, or a body temperature>38℃)
10. Significant peripheral arterial disease affecting the upper limbs
11. surgeries: cardiac transplantation, concomitant carotid endarterectomy , previous heart surgery,, off-pump surgery, emergency surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-02-07 (Actual); Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of PaO2/FiO2 over 24 hours after cardiac surgery | 24 hours post surgery

SECONDARY OUTCOMES:
All-cause mortality | 30 days post surgery
Postoperative Pulmonary Complications | 30 days post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Liu Su, M.D/Ph.D, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
IPD will be available when this trial is finished and the article have been published.

REFERENCES:
- [Result] Domanski MJ, Mahaffey K, Hasselblad V, Brener SJ, Smith PK, Hillis G, Engoren M, Alexander JH, Levy JH, Chaitman BR, Broderick S, Mack MJ, Pieper KS, Farkouh ME. Association of myocardial enzyme elevation and survival following coronary artery bypass graft surgery. JAMA. 2011 Feb 9;305(6):585-91. doi: 10.1001/jama.2011.99. PMID 21304084
- [Result] JENNINGS RB, SOMMERS HM, SMYTH GA, FLACK HA, LINN H. Myocardial necrosis induced by temporary occlusion of a coronary artery in the dog. Arch Pathol. 1960 Jul;70:68-78. No abstract available. PMID 14407094
- [Result] Braunwald E, Kloner RA. Myocardial reperfusion: a double-edged sword? J Clin Invest. 1985 Nov;76(5):1713-9. doi: 10.1172/JCI112160. No abstract available. PMID 4056048
- [Result] Sullivan PJ, Sweeney KJ, Hirpara KM, Malone CB, Curtin W, Kerin MJ. Cyclical ischaemic preconditioning modulates the adaptive immune response in human limb ischaemia-reperfusion injury. Br J Surg. 2009 Apr;96(4):381-90. doi: 10.1002/bjs.6554. PMID 19283744
- [Result] Bolli R. The late phase of preconditioning. Circ Res. 2000 Nov 24;87(11):972-83. doi: 10.1161/01.res.87.11.972. PMID 11090541
- [Result] Murry CE, Jennings RB, Reimer KA. Preconditioning with ischemia: a delay of lethal cell injury in ischemic myocardium. Circulation. 1986 Nov;74(5):1124-36. doi: 10.1161/01.cir.74.5.1124. PMID 3769170
- [Result] Przyklenk K, Bauer B, Ovize M, Kloner RA, Whittaker P. Regional ischemic 'preconditioning' protects remote virgin myocardium from subsequent sustained coronary occlusion. Circulation. 1993 Mar;87(3):893-9. doi: 10.1161/01.cir.87.3.893. PMID 7680290
- [Result] Gho BC, Schoemaker RG, van den Doel MA, Duncker DJ, Verdouw PD. Myocardial protection by brief ischemia in noncardiac tissue. Circulation. 1996 Nov 1;94(9):2193-200. doi: 10.1161/01.cir.94.9.2193. PMID 8901671
- [Result] Oxman T, Arad M, Klein R, Avazov N, Rabinowitz B. Limb ischemia preconditions the heart against reperfusion tachyarrhythmia. Am J Physiol. 1997 Oct;273(4):H1707-12. doi: 10.1152/ajpheart.1997.273.4.H1707. PMID 9362234
- [Result] Li G, Labruto F, Sirsjo A, Chen F, Vaage J, Valen G. Myocardial protection by remote preconditioning: the role of nuclear factor kappa-B p105 and inducible nitric oxide synthase. Eur J Cardiothorac Surg. 2004 Nov;26(5):968-73. doi: 10.1016/j.ejcts.2004.06.015. PMID 15519191
- [Result] Kharbanda RK, Mortensen UM, White PA, Kristiansen SB, Schmidt MR, Hoschtitzky JA, Vogel M, Sorensen K, Redington AN, MacAllister R. Transient limb ischemia induces remote ischemic preconditioning in vivo. Circulation. 2002 Dec 3;106(23):2881-3. doi: 10.1161/01.cir.0000043806.51912.9b. PMID 12460865
- [Result] Hausenloy DJ, Yellon DM. Remote ischaemic preconditioning: underlying mechanisms and clinical application. Cardiovasc Res. 2008 Aug 1;79(3):377-86. doi: 10.1093/cvr/cvn114. Epub 2008 May 2. PMID 18456674
- [Result] Sivaraman V, Pickard JM, Hausenloy DJ. Remote ischaemic conditioning: cardiac protection from afar. Anaesthesia. 2015 Jun;70(6):732-48. doi: 10.1111/anae.12973. Epub 2015 Feb 26. PMID 25961420
- [Result] Heusch G, Botker HE, Przyklenk K, Redington A, Yellon D. Remote ischemic conditioning. J Am Coll Cardiol. 2015 Jan 20;65(2):177-95. doi: 10.1016/j.jacc.2014.10.031. PMID 25593060
- [Result] Kerendi F, Kin H, Halkos ME, Jiang R, Zatta AJ, Zhao ZQ, Guyton RA, Vinten-Johansen J. Remote postconditioning. Brief renal ischemia and reperfusion applied before coronary artery reperfusion reduces myocardial infarct size via endogenous activation of adenosine receptors. Basic Res Cardiol. 2005 Sep;100(5):404-12. doi: 10.1007/s00395-005-0539-2. Epub 2005 Jun 17. PMID 15965583
- [Result] Hausenloy DJ, Mwamure PK, Venugopal V, Harris J, Barnard M, Grundy E, Ashley E, Vichare S, Di Salvo C, Kolvekar S, Hayward M, Keogh B, MacAllister RJ, Yellon DM. Effect of remote ischaemic preconditioning on myocardial injury in patients undergoing coronary artery bypass graft surgery: a randomised controlled trial. Lancet. 2007 Aug 18;370(9587):575-9. doi: 10.1016/S0140-6736(07)61296-3. PMID 17707752
- [Result] Hammermeister KE, Burchfiel C, Johnson R, Grover FL. Identification of patients at greatest risk for developing major complications at cardiac surgery. Circulation. 1990 Nov;82(5 Suppl):IV380-9. PMID 2225429
- [Result] Messent M, Sullivan K, Keogh BF, Morgan CJ, Evans TW. Adult respiratory distress syndrome following cardiopulmonary bypass: incidence and prediction. Anaesthesia. 1992 Mar;47(3):267-8. doi: 10.1111/j.1365-2044.1992.tb02134.x. PMID 1566999
- [Result] Wan S, LeClerc JL, Vincent JL. Inflammatory response to cardiopulmonary bypass: mechanisms involved and possible therapeutic strategies. Chest. 1997 Sep;112(3):676-92. doi: 10.1378/chest.112.3.676. PMID 9315800
- [Result] Kharbanda RK, Li J, Konstantinov IE, Cheung MM, White PA, Frndova H, Stokoe J, Cox P, Vogel M, Van Arsdell G, MacAllister R, Redington AN. Remote ischaemic preconditioning protects against cardiopulmonary bypass-induced tissue injury: a preclinical study. Heart. 2006 Oct;92(10):1506-11. doi: 10.1136/hrt.2004.042366. Epub 2006 Jul 3. PMID 16818489
- [Result] Xia Z, Herijgers P, Nishida T, Ozaki S, Wouters P, Flameng W. Remote preconditioning lessens the deterioration of pulmonary function after repeated coronary artery occlusion and reperfusion in sheep. Can J Anaesth. 2003 May;50(5):481-8. doi: 10.1007/BF03021061. English, French. PMID 12734158
- [Result] Cheung MM, Kharbanda RK, Konstantinov IE, Shimizu M, Frndova H, Li J, Holtby HM, Cox PN, Smallhorn JF, Van Arsdell GS, Redington AN. Randomized controlled trial of the effects of remote ischemic preconditioning on children undergoing cardiac surgery: first clinical application in humans. J Am Coll Cardiol. 2006 Jun 6;47(11):2277-82. doi: 10.1016/j.jacc.2006.01.066. Epub 2006 May 15. PMID 16750696
- [Result] Zhou W, Zeng D, Chen R, Liu J, Yang G, Liu P, Zhou X. Limb ischemic preconditioning reduces heart and lung injury after an open heart operation in infants. Pediatr Cardiol. 2010 Jan;31(1):22-9. doi: 10.1007/s00246-009-9536-9. Epub 2009 Sep 29. PMID 19787388
- [Result] Kim JC, Shim JK, Lee S, Yoo YC, Yang SY, Kwak YL. Effect of combined remote ischemic preconditioning and postconditioning on pulmonary function in valvular heart surgery. Chest. 2012 Aug;142(2):467-475. doi: 10.1378/chest.11-2246. PMID 22281799
- [Result] Li L, Luo W, Huang L, Zhang W, Gao Y, Jiang H, Zhang C, Long L, Chen S. Remote perconditioning reduces myocardial injury in adult valve replacement: a randomized controlled trial. J Surg Res. 2010 Nov;164(1):e21-6. doi: 10.1016/j.jss.2010.06.016. Epub 2010 Jul 2. PMID 20850778
- [Result] Rahman IA, Mascaro JG, Steeds RP, Frenneaux MP, Nightingale P, Gosling P, Townsend P, Townend JN, Green D, Bonser RS. Remote ischemic preconditioning in human coronary artery bypass surgery: from promise to disappointment? Circulation. 2010 Sep 14;122(11 Suppl):S53-9. doi: 10.1161/CIRCULATIONAHA.109.926667. PMID 20837926